CLINICAL TRIAL: NCT02752464
Title: Behavioral Cardiovascular Disease Prevention Using Informatics
Brief Title: Behavioral CVD Prevention Using Informatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Lisa M. Quintiliani, Assistant Professor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-34964; 14SDG20050015 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Health Behavior
Keywords: Weight Loss; Health Status Disparities
MeSH Terms: conditions — Health Behavior; Weight Loss | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback report plus peer counseling (Experimental): Feedback report plus peer counseling Participants receive 12 sessions of behavioral counseling and a brief printed feedback report
  Interventions: Behavioral: Counseling; Behavioral: feedback report
- Feedback report (Active Comparator): Feedback report Participants receive a brief printed feedback report
  Interventions: Behavioral: feedback report

INTERVENTIONS:
Behavioral: Counseling — Up to 12 sessions of behavioral counseling using motivational interviewing techniques focused on diet and physical activity behaviors over a 12 week period. Counselors will be guided in their sessions by a computer program called CuesWeight. Participants also receive text messages to enable participants to track their behaviors; this information is relayed to the counselors to inform the counseling sessions.
  Arms: Feedback report plus peer counseling
Behavioral: feedback report — All participants receive a brief printed feedback report displaying their current levels of nutrition and physical activity behaviors and tips for meeting recommended guidelines.

SUMMARY:
Overweight/obesity is strongly linked to mortality from multiple chronic diseases, including cardiovascular disease, diabetes, and obesity-related cancers.The successful management of overweight/obesity requires management of nutrition and physical activity over time. For racial/ethnic minority and low-income populations, who face both higher prevalence of obesity and chronic diseases compared to others, interventions promoting behavioral change are a national health priority. From the available range of behavioral change intervention strategies, there is a growing knowledge base that documents the efficacy of peer support interventions for improving self-care, quality of life, and behavioral change. In this study, the investigators will examine the following research question: What is the preliminary efficacy and degree of implementation and acceptability of an intervention approach in which peer counselors provide evidenced-based counseling about nutrition and physical activity behaviors for weight management to public housing residents using a computer-assisted program called CuesWeight?

ELIGIBILITY:
Inclusion Criteria:

* Willing to wear an accelerometer
* 18-65 years old
* Public housing resident with no plans to move in next 6 months
* Body mass index ≥25
* Open to making changes to diet & physical activity habits

Exclusion Criteria:

* Currently enrolled in a comprehensive weight loss program or a research study whose primary outcome is weight loss
* Primary language spoken is a language other than Spanish or English
* Not willing to participate in study protocols, including wearing the accelerometer, not willing to have study staff send text messages

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Weight-objective measurement | 12 weeks
  Weight in pounds will be measured objectively with a digital scale

SECONDARY OUTCOMES:
Diet, fruits and vegetables, self-reported via questionnaire | 12 weeks
  Servings of fruits and vegetables will be measured via the Primescreen dietary screener instrument
Diet, sugar sweetened beverages, self-reported via questionnaire | 12 weeks
  Fluid ounces of sugar sweetened beverages will be measured via the BEV-Q questionnaire
Diet, fast food, self-reported via questionnaire | 12 weeks
  Number of visits to fast food restaurants will be measured via a 1-item question asking participants how often they go to fast food restaurants
Physical activity, objectively measured | 12 weeks
  Minutes of light to moderate physical activity will be measured via accelerometers (Actigraphs)
Physical activity, self-reported | 12 weeks
  Minutes of light to moderate physical activity will be measured via a questionnaire (IPAQ)
Internal motivation, self-reported via questionnaire | 12 weeks
  Perceptions of internal motivation to change diet and physical activity will be measured by a brief questionnaire
Self-efficacy for eating a healthful diet, self-reported via questionnaire | 12 weeks
  Perceptions of self-efficacy (or confidence) to change diet behaviors in a variety of situations will be measured by a brief questionnaire
Self-efficacy for doing physical activity, self-reported via questionnaire | 12 weeks
  Perceptions of self-efficacy (or confidence) to change physical activity behaviors in a variety of situations will be measured by a brief questionnaire
Social support, self-reported via questionnaire | 12 weeks
  Perceptions of social support from a variety of sources will be measured via a brief questionnaire
Feasibility, number of counseling sessions completed | 12 weeks
  Number of counseling sessions completed in-person and over the phone will be tallied and reported
Feasibility, acceptability of intervention | 12 weeks
  Perceptions of acceptability of both the brief feedback report and the counseling sessions will be asked in open- and closed-ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Quintiliani, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No